CLINICAL TRIAL: NCT01481805
Title: Biomarker Analysis in Sorafenib Treated Hepatocellular Carcinoma Patients
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ho Yeong Lim, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Other Study IDs: 2009-09-055
Record Dates: First submitted 2011-11-16; First posted 2011-11-30 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatocellular carcinoma patients treated with sorafenib

SUMMARY:
To explore biomarkers predictive of clinical response to sorafenib in unresectable hepatocellular carcinoma using the Prometheus Platform To analyze expression and activation status of receptor tyrosine kinases in signal transduction pathways in FNA samples and circulating tumor cells.

To identify negative predictive markers to sorafenib. To elucidate signal transduction pathway attributable to sorafenib resistance. To monitor changes in the RTK activation status during sorafenib treatment using circulating tumor cells.

To analyze correlation between the quantity of circulating tumor cells and circulating endothelial cell precursors and treatment response to sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed hepatocellular carcinoma (HCC) or a combination of radiologically compatible finding to HCC, alpha-fetoprotein > 400ng/mL and liver cirrhosis
* Inoperable disease as defined by (Localized disease in a portion of the liver that doses not allow the possibility of complete surgical removal of the tumor with a clear resection margin OR Presence of extra-hepatic disease OR Main portal vein or hepatic vein involvement (invasion or tumor thrombus) OR The HCC must not be amenable to intra-arterial therapy or local ablative therapy)
* Minimum life expectancy of 12 weeks
* Age > 18 years.
* ECOG Performance Status of ≤ 2
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

(Hemoglobin > 9.0 g/dl,Absolute neutrophil count>1,500/mm3, Platelet count>75,000/μl,Total bilirubin < 1.5 times the upper limit of normal,ALT and AST < 5 x upper limit of normal,Albumin ≥ 3g/dL,PT-INR/PTT < 1.5 x upper limit of normal,Serum creatinine < 1.5 x upper limit of normal or Creatinine clearance ≥ 50mL/min)

* Signed and dated informed consent before the start of specific protocol procedures.
* FNA will be performed in patients with feasible biopsy site

Exclusion Criteria:

* Decompensated cirrhosis or stage C (Index > 10) according to the Child-Pugh Classification
* Other concomitant anticancer agent, including Tamoxifen and Interferon
* Active clinically serious infections (> grade 2 CTCAE version 3.0)
* History of organ allograft
* Patients with evidence or history of bleeding diasthesis
* Patients undergoing renal dialysis
* Radiotherapy during study or within 4 weeks of start of study drug.
* Prior exposure to the study drug.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatocellular carcinoma patients treated with sorafenib
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-01-14 (Actual); Primary Completion 2014-01-13 (Actual); Study Completion 2014-08-13 (Actual)

PRIMARY OUTCOMES:
Biomarkers predictive | 36months
  To explore biomarkers predictive of clinical response to sorafenib in unresectable hepatocellular carcinoma using the Prometheus Platform A. To analyze expression and activation status of receptor tyrosine kinases in signal transduction pathways in FNA samples and circulating tumor cells B. To identify negative predictive markers to sorafenib

SECONDARY OUTCOMES:
Signal transduction pathway | 36months
  To elucidate signal transduction pathway attributable to sorafenib resistance.
The RTK activation status. | 36months
  To monitor changes in the RTK activation status during sorafenib treatment using circulating tumor cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical Center, Seoul, South Korea